CLINICAL TRIAL: NCT05210517
Title: Uric Acid Excretion Study: Open-label Randomised Cross Over Study
Brief Title: SGLT2 Inhibition: Uric Acid Excretion Study
Acronym: UREX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, D van Raalte, MD PhD, associate professor of medicine, internist-endocrinologist, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DCUREX2021
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Benzbromarone

STUDY DESIGN:
Intervention Model Description: 4-arm cross over, open label intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No intervention (No Intervention)
- Empagliflozin (Experimental): Empagliflozin 25 mg once daily for one week
  Interventions: Drug: Empagliflozin 25 MG
- Benzbromarone (Experimental): Benzbromarone 100 mg once daily for one week
  Interventions: Drug: Benzbromaron
- Empagliflozin-Benzbromarone (Experimental): Empagliflozin 25 mg once daily for one week combined with Benzbromarone 100 mg once daily for one week
  Interventions: Drug: Empagliflozin 25 MG + benzbromarone 100 mg

INTERVENTIONS:
Drug: Empagliflozin 25 MG — 25 once daily one week treatment
  Arms: Empagliflozin
Drug: Benzbromaron — 100 mg once daily 1 one week treatment
  Arms: Benzbromarone
Drug: Empagliflozin 25 MG + benzbromarone 100 mg — combined treatment once daily for one week
  Arms: Empagliflozin-Benzbromarone

SUMMARY:
The current study investigates the effects of SGLT2 inhibitor empagliflozin on uric acid excretion.

DETAILED DESCRIPTION:
SGTL2 inhibitors improve cardiovascular and kidney outcomes. The underlying mechanisms are incompletely understood. SGLT2 inhibitors are known to reduce plasma uric acid likely by enhanced urinary uric acid excretion.

In this study the investigators will study the effects of SGLT2 inhibit on uric acid levels and excretion in detail, linking it to the role of glucosuria and Uric acid transporter (URAT1) which in rodents was indispensable for the glucose-lowering effects of SGLT2 inhibition.

ELIGIBILITY:
Inclusion Criteria:

Caucasian Men or post-menopausal women Age 35 to 75 Diagnosed with T2D HbA1c from 6.5% to 9.0% (48-75 mmol/mol) body mass index >25 kg/m2 Treated with metformin monotherapy (stable dose for ≥3 months) with or without sulfonylurea Well-controlled blood pressure (i.e., <140/90 mm Hg). In case of previously diagnosed hypertension and/or albuminuria treatment at least a stable dose of a renin-angiotensin system (RAS) inhibitor for ≥3 months at maximal tolerable dose.

Exclusion Criteria:

History of gout history of unstable or rapidly progressing renal or malignant disease (excluding basal cell carcinoma) eGFR <60 mL/min/1.73 m2 Estimated GFR <45 mL/min/1.73m2 (determined by the Modification of Diet in Renal Disease (MDRD) study equation) Hemoglobin level < 7.0 mmol/L Current urinary tract infection and active nephritis Macroalbuminuria; defined as ACR of >300 mg/g. Current/chronic use of the following medication: thiazolidinediones, sulfonylurea derivatives, GLP-1 receptor agonists, DPP-4 inhibitors, SGLT-2 inhibitor, oral glucocorticoids, immune suppressants, antimicrobial agents, chemotherapeutics, antipsychotics, tricyclic antidepressants (TCAs) and monoamine oxidase inhibitors (MOAIs).

Patients on diuretics will only be excluded when these drugs cannot be stopped 3 months prior randomization and for the duration of the study.

Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs) will not be allowed, unless used as incidental medication (1-2 tablets) for non-chronic indications (i.e. sports injury, head-ache or back ache). However, no such drugs can be taken within a time-frame of 2 weeks prior to renal-testing Pregnancy History of or actual severe mental disease History of or actual severe somatic disease (e.g. systemic disease) History of or actual malignancy (except basal cell carcinoma) History of or actual pancreatic disease (Unstable) thyroid disease Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) Recent (<6 months) history of cardiovascular disease, including Acute coronary syndrome Stroke or transient ischemic neurologic disorder or chronic heart failure (NYHA grade II-IV) Complaints compatible with or established neurogenic bladder and/or incomplete bladder emptying (as determined by ultrasonic bladder scan) Substance abuse (alcohol: defined as >3 units alcohol/day) History of diabetic ketoacidosis (DKA) requiring medical intervention (e.g., emergency room visit and/or hospitalization) within 1 month prior to the Screening visit.

Recent blood donation (< 6 months) Allergy to any of the agents used in the study Inability to understand the protocol and/or give informed consent Individuals who are investigator site personnel, directly affiliated with the study, or are immediate (spouse, parent, child, or sibling, whether biological or legally adopted) family of investigator site personnel directly affiliated with the study

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
plasma uric acid | 1 week
  change in plasma uric acid concentrations
Fractional uric acid excretion | one week
  change creatinine-adjusted fractional uric acid excretion

SECONDARY OUTCOMES:
urinary glucose levels | one week
  glucose concentration urine

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suijk DLS, van Baar MJB, van Bommel EJM, Iqbal Z, Krebber MM, Vallon V, Touw D, Hoorn EJ, Nieuwdorp M, Kramer MMH, Joles JA, Bjornstad P, van Raalte DH. SGLT2 Inhibition and Uric Acid Excretion in Patients with Type 2 Diabetes and Normal Kidney Function. Clin J Am Soc Nephrol. 2022 May;17(5):663-671. doi: 10.2215/CJN.11480821. Epub 2022 Mar 23. PMID 35322793